CLINICAL TRIAL: NCT05657704
Title: Randomized Clinical Trial to Evaluate the Utility of CYP2D6 Genotyping to Improve the Efficacy and Safety of Tramadol in the Treatment of Acute Postoperative Pain.
Brief Title: Utility of CYP2D6 Genotyping to Improve the Efficacy and Safety of Tramadol
Acronym: Tradol-PriME
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Hospital Universitario La Paz (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Fundación Jiménez Díaz (Other); Hospital Universitario San Juan de Alicante (Other); Hospital Universitario de Burgos (Other); Hospital San Carlos, Madrid (Other); Puerta de Hierro University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-500377-13-01
Record Dates: First submitted 2022-10-10; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Post-surgical Pain; Pain, Acute; Postoperative Pain
Keywords: Pharmacogenetics; Therapeutic techniques in treatment of acute postoperative pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Tramadol; dexketoprofen trometamol

STUDY DESIGN:
Intervention Model Description: Phase IV trial and low intervention, multicenter study. Group 1: Tramadol, 100 mg according to clinical practice for the treatment of postoperative pain. Group 2: Dexketoprofen 25 mg according to clinical practice for the treatment of postoperative pain. Experimental group 3: patients in this group will be genotyped before surgery and treatment will be prescribed according to the CYP2D6 phenotype. Normal Metabolizers (NM): Tramadol 100 mg every 8 hour; Ultrarapid Metabolizers (UM): Tramadol 50 mg every 8 hours and Intermediate and poor metabolizers (IM/PM): dexketoprofen 25 mg every 8 hours
Masking Description: Open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tramadol (No Intervention): Patients treated with Tramadol, 100 mg every 8 hours according to clinical practice for the treatment of postoperative pain.
- Dexketoprofen (No Intervention): Patients treated with Dexketoprofen 25 mg every 8 hours according to clinical practice for the treatment of postoperative pain.
- Experimental Group (Experimental): The patients in this group will be genotyped before surgery and treatment will be prescribed according to the CYP2D6 phenotype.
  Normal Metabolizers (NM): Tramadol 100 mg every 8 hour; Ultrarapid Metabolizers (UM): Tramadol 50 mg every 8 hours Intermediate and poor metabolizers (IM/PM): dexketoprofen 25 mg every 8 hours
  Interventions: Drug: The patients in experimental group will be genotyped before surgery and treatment will be prescribed according to the CYP2D6 phenotype

INTERVENTIONS:
Drug: The patients in experimental group will be genotyped before surgery and treatment will be prescribed according to the CYP2D6 phenotype — Treatment will be prescribed according to the CYP2D6 phenotype. Normal Metabolizers (NM): Tramadol 100 mg every 8 hour; Ultrarapid Metabolizers (UM): Tramadol 50 mg every 8 hours Intermediate and poor metabolizers (IM/PM): dexketoprofen 25 mg every 8 hours
  Other Names: Tramadol 100 mg; Tramadol 50 mg; Dexketoprofen 25 mg
  Arms: Experimental Group

SUMMARY:
Randomized clinical trial to evaluate the utility of CYP2D6 genotyping to improve the efficacy and safety of tramadol in the treatment of acute postoperative pain.

Phase IV and low-intervention trial To evaluate if the implementation of pharmacogenetics in clinical practice can help to improve the treatment of acute pain, increasing efficacy and reducing adverse reactions.

The main evaluation variable: This is a simple study, which does not differ from standard clinical practice and therefore we do not expect early ending of the study.

DETAILED DESCRIPTION:
Randomized clinical trial to evaluate the utility of CYP2D6 genotyping to improve the efficacy and safety of tramadol in the treatment of acute postoperative pain.

Phase IV and low-intervention trial The main objective is evaluate if the implementation of pharmacogenetics in clinical practice can help to improve the treatment of acute pain, increasing efficacy and reducing adverse reactions. Secondary objectives: 1. To evaluate whether treatment adjusted according to CYP2D6 phenotype can reduce adverse reactions to tramadol in acute postoperative pain. 2. To compare the efficacy and safety of dexketoprofen and tramadol in the treatment of acute postoperative pain. 3. To investigate the influence on analgesic response and the incidence of adverse reactions of polymorphisms of other genes involved in the pharmacokinetics and mechanism of action of dexketoprofen and tramadol, such as: CYP2C9, CYP2C8, CYP2C19, CYP3A4, CYP3A5, CYP2B6, CYP2E1, COMT, ABCB1, SLC22A1, OPRM1 and PTGS2. 4. To evaluate the relationship of tramadol, M1 and dexketoprofen plasma concentrations with response to treatment and the occurrence of adverse reactions.

Inclusion criteria: 1. Men or women over 18 years of age. 2. Patients scheduled for outpatient surgical extraction, under local anesthesia, of at least two impacted third molars, at least one of which will require bone removal. 3. Patients who agree to participate in the study and give written consent.

Exclusion criteria: 1. Patients under treatment with other drugs that can inhibit CYP2D6, or are contraindicated in combination with tramadol or dexketoprofen. 2. Patients on treatment with bisphosphonates. 3. Patients who are receiving analgesic treatment before the operation, 24 hours prior to the operation. This criterion will be evaluated at the intervention visit. 4. Patients suffering from other uncontrolled diseases. 5. Pregnant or breastfeeding women. 6. Patients with contraindications for treatment with tramadol or dexketoprofen.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years of age.
* Patients scheduled for outpatient surgical extraction, under local anesthesia, of at least two impacted third molars, at least one of which will require bone removal.
* Patients who agree to participate in the study and give written consent.

Exclusion Criteria:

* Patients under treatment with other drugs that can inhibit CYP2D6, or are contraindicated in combination with tramadol or dexketoprofen.
* Patients on treatment with bisphosphonates.
* Patients who are receiving analgesic treatment before the operation, 24 hours prior to the operation. This criterion will be evaluated at the intervention visit.
* Patients suffering from other uncontrolled diseases.
* Pregnant or breastfeeding women.
* Patients with contraindications for treatment with tramadol or dexketoprofen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy: analgesic effect (Pain assessment) 4 hours after treatment | 4 hour after treatment
  To evaluate the analgesic effect (pain assessment) that will be evaluated throughout visual analogical scale (VAS) from 0 to 100.

SECONDARY OUTCOMES:
Efficacy at the end of treatment | 3 days after treatment administration (72 Hours)
  Efficacy will also be evaluated based on the requirement of the study medication, if treatment has been completed during the three days (recommended in the study protocol), or on the contrary, three days of treatment have not been required due to pain remission; the requirement of rescue medication due to lack of efficacy of the prescribed treatments in the first 24 hours after the administration of the first dose. Time to rescue medication use will also be measured.
Correlation between efficacy and the pharmacokinetic parameters (AUC) | 1 hours, 2 hours and 4 hours
  The efficacy of the treatments will be analyzed and whether these correlate with the pharmacokinetic parameters (AUC) for each patient, calculated from the quantified plasma concentrations of tramadol and metabolite1 of tramadol (samples 2 hour and 4h) or dexketoprofen (samples 1h and 4h).
Correlation between efficacy and pharmacogenetic profile (focus in CYP2D6) | Through study completion, an average of 1 year and 6 months
  The efficacy of the treatments will be analyzed with the pharmacogenetic profile of the patients, that is, if the pharmacokinetic profile, Tmax and AUC, correlates with the enzymatic activity rate for the CYP2D6 phenotype (Activity Score - AS) of poor metabolizer (AS-0), intermediate metabolizer (AS: between 0 and 1.25), normal metabolizer ( AS: between 1.25 and 2.25) or ultrarapid metabolizer (AS > 2.25)
Safety evaluations | Through study completion, an average of 1 year and 6 months
  The safety evaluations will be carried out in accordance with the Good Clinical Practice Standards and current legislation. The safety of the treatments will be analyzed with the pharmacogenetic profile of the patients

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (8):
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario San Juan de Alicante, Alicante
  - Hospital General Universitario de Burgos y Clínica Colina, Burgos
  - Fundación para la Investigación Biomédica Hospital La Princesa, Madrid
  - Hospital Univesitario Ramón y Cajal, Madrid
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hostpital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitaro La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No